CLINICAL TRIAL: NCT00981422
Title: Search for Biomarkers in Human Glaucoma: Possible Correlations Between Alterations in Peripheral Lymphocytes and Disease Severity
Brief Title: Search for Biomarkers in Human Glaucoma: Lymphocytes Alterations and Rate of Progression
Status: Completed | Type: Observational
Sponsor: University of Parma (Other)
Responsible Party: STEFANO GANDOLFI, Professor of Ophthalmology and Chairman, UNIVERSITY OF PARMA
Other Study IDs: PARMABIOMARKERS001
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Glaucoma, Open-Angle
Keywords: glaucoma; immunology; immunophenotype
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Glaucoma patients: POAG patients selected by an ophthalmologist from the Glaucoma Service, Ophthalmology Institute, University of Parma
- Healthy: healthy subjects with negative history for (a) neurodegenerative diseases, (b) autoimmune diseases, (c) cancer, (d) viral infection, (e) diabetes, and (f) systemic inflammation

SUMMARY:
The aim of this study was to evaluate the lymphocyte phenotype in primary open- angle glaucoma (POAG) patients compared to healthy subjects of the same age, in order to confirm the importance of immune responses in glaucoma and the possible correlation to the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary open-angle glaucoma
* age between 19 an 85 years old

Exclusion Criteria:

* age less than 19 or more than 85 yrs
* positive history for (a) neurodegenerative diseases, (b) autoimmune diseases, (c) cancer, (d) viral infection and (e) diabetes, (f)systemic inflammation

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic in Parma (University hospital of Parma)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
compare the lymphocyte phenotype of POAG patients to healthy subjects of the same age | the same day of bloodwithdrawal

SECONDARY OUTCOMES:
correlate the immunophenotype of POAG patients to the severity of disease | within 3 months after blood withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Stefano A Gandolfi, MD, Principal Investigator — Ophthalmology Institute, University of Parma, Italy
Locations (1):
- Azienda ospedaliera universitaria, Parma, Italy